CLINICAL TRIAL: NCT01615029
Title: An Open Label, International, Multicenter, Dose Escalating Phase I/II Trial Investigating the Safety of Daratumumab in Combination With Lenalidomide and Dexamethasone in Patients With Relapsed or Relapsed and Refractory Multiple Myeloma
Brief Title: Daratumumab in Combination With Lenalidomide and Dexamethasone in Relapsed and Relapsed-refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR101391; DARA-GEN503 (Other: Janssen Research & Development, LLC); 2011-005709-62 (EudraCT Number)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Daratumumab; Lenalidomide; Dexamethasone; Dose-escalation; Relapsed multiple myeloma; Relapsed and refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Daratumumab (Experimental): Participants will receive daratumumab along with Lenalidomide and dexamethasone.
  Interventions: Drug: Part 1 (Dose Escalation): Daratumumab; Drug: Part 2 (Dose Expansion): Daratumumab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Part 1 (Dose Escalation): Daratumumab — Participants will receive intravenous (injection of a substance into a vein) infusion of daratumumab in an increased fashion from 2 milligram per kilogram (mg/kg) up to maximum dose of 16 mg/kg. Considering the safety and efficacy of dose in Part 1, recommended phase 2 dose (RP2D) for Part 2 of the study will be decided. A predose infusion of 10 percent (%) of the full dose of daratumumab will be administered a day before the first full infusion of the first cycle. Participants will receive 4 weekly infusions in the first 2 treatment cycles. From cycles 3 to 6 infusions will be administered every alternate week and monthly infusions will be administered from cycle 7 until disease progression.
Drug: Part 2 (Dose Expansion): Daratumumab — Participants will receive RP2D as determined in Part 1 of the study. Participants will receive 4 weekly infusions of RP2D in the first 2 treatment cycles. From cycles 3 to 6 infusions will be administered every alternate week and monthly infusions will be administered from cycle 7 until disease progression.
Drug: Lenalidomide — All participants (Part 1 and Part 2) will receive 25 mg lenalidomide orally (by mouth) from days 1 to 21 of each 28-day cycle until disease progression.
Drug: Dexamethasone — All participants (Part 1 and Part 2) will receive 40 mg (20 mg intravenously [injection of a substance into a vein]) dexamethasone once weekly. Participants older than 75 years or underweight (body mass index [BMI] less than [<] 18.5), the dexamethasone dose will be administered at a dose of 20 mg once weekly until disease progression.

SUMMARY:
The purpose of this study is to establish the safety profile of daratumumab when given in combination with Lenalidomide and dexamethasone in participants with relapsed or relapsed and refractory Multiple Myeloma (MM).

DETAILED DESCRIPTION:
The study is conducted in two parts. The dose escalation portion of the trial (Part 1) participants are enrolled into cohorts at increasing dose levels of daratumumab in combination with Len/Dex in 28 day treatment cycles. Part 2, the cohort expansion part of the trial, will further explore the maximum tolerated dose (MTD) (or the maximum tested dose) of daratumumab as determined in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* (Part 1) Have relapsed multiple myeloma after receiving a minimum of 2 and a maximum of 4 prior lines of therapy and be eligible for treatment with lenalidomide and dexamethasone (Len/Dex)
* (Part 2) Have received at least 1 prior line of therapy for multiple myeloma
* Be older than or be 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status (0-2)
* Provide signed informed consent after receipt of oral and written information about the study and before any study-related activity is performed

Exclusion Criteria:

* Have previously received an allogenic stem cell transplant
* Have received autologous stem cell transplant within 12 weeks before the first infusion
* Have received antimyeloma treatment, radiotherapy, or any experimental drug or therapy within 2 weeks before the first infusion
* Have discontinued lenalidomide due to any treatment-related adverse event or be refractory to any dose of lenalidomide. Refractory to lenalidomide is defined as either, participants whose disease progresses within 60 days of lenalidomide, or participants whose disease is nonresponsive while on any dose of lenalidomide. Nonresponsive disease is defined as either failure to achieve at least an minimal response (MR) or development of progressive disease (PD) while on lenalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-06-26 (Actual); Primary Completion 2015-10-02 (Actual); Study Completion 2024-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC; Torben Plesner, MD, Principal Investigator — Vejle Hospital; Paul Richardson, MD, Principal Investigator — Dana Farber
Locations (8):
- Boston, Massachusetts, United States
- Denmark (2):
  - Copenhagen Ø
  - Vejle
- France (3):
  - Lille
  - Nantes
  - Vandœuvre-lès-Nancy
- Utrecht, Netherlands
- London, United Kingdom

REFERENCES:
- [Derived] Krejcik J, Frerichs KA, Nijhof IS, van Kessel B, van Velzen JF, Bloem AC, Broekmans MEC, Zweegman S, van Meerloo J, Musters RJP, Poddighe PJ, Groen RWJ, Chiu C, Plesner T, Lokhorst HM, Sasser AK, Mutis T, van de Donk NWCJ. Monocytes and Granulocytes Reduce CD38 Expression Levels on Myeloma Cells in Patients Treated with Daratumumab. Clin Cancer Res. 2017 Dec 15;23(24):7498-7511. doi: 10.1158/1078-0432.CCR-17-2027. Epub 2017 Oct 12. PMID 29025767
- [Derived] Plesner T, Arkenau HT, Gimsing P, Krejcik J, Lemech C, Minnema MC, Lassen U, Laubach JP, Palumbo A, Lisby S, Basse L, Wang J, Sasser AK, Guckert ME, de Boer C, Khokhar NZ, Yeh H, Clemens PL, Ahmadi T, Lokhorst HM, Richardson PG. Phase 1/2 study of daratumumab, lenalidomide, and dexamethasone for relapsed multiple myeloma. Blood. 2016 Oct 6;128(14):1821-1828. doi: 10.1182/blood-2016-07-726729. Epub 2016 Aug 16. PMID 27531679

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: 2 mg/kg Daratumumab + Lenalidomide and Dexamethasone: Participants administered with daratumumab 2 milligram/kilogram (mg/kg) on Day 0 (pre dose infusion), 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Days 1 and 15 (Cycles 3 to 6), Day 1 (Cycle 7+) along with Lenalidomide 25 milligram (mg) on Day 1 to 21 of each 28-day cycle and Dexamethasone 40 mg (weekly) and may be reduced to 20 mg (weekly after cycle 6 at the investigator's discretion). Each treatment cycle consists of 28 days.
- Phase 1: 4 mg/kg Daratumumab + Lenalidomide and Dexamethasone: Participants administered with daratumumab 4 mg/kg on Day 0 (pre dose infusion), 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Days 1 and 15 (Cycles 3 to 6), Day 1 (Cycle 7+) along with Lenalidomide 25 mg on Day 1 to 21 of each 28-day cycle and Dexamethasone 40 mg (weekly) and may be reduced to 20 mg (weekly after cycle 6 at the investigator's discretion). Each treatment cycle consists of 28 days.
- Phase 1: 8mg/kg Daratumumab + Lenalidomide and Dexamethasone: Participants administered with daratumumab 8 mg/kg on Day 0 (pre dose infusion), 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Days 1 and 15 (Cycles 3 to 6), Day 1 (Cycle 7+) along with Lenalidomide 25 mg on Day 1 to 21 of each 28-day cycle and Dexamethasone 40 mg (weekly) and may be reduced to 20 mg (weekly after cycle 6 at the investigator's discretion). Each treatment cycle consists of 28 days.
- Phase 1: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone: Participants administered with daratumumab 16 mg/kg on Day 0 (pre dose infusion), 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Days 1 and 15 (Cycles 3 to 6), Day 1 (Cycle 7+) along with Lenalidomide 25 mg on Day 1 to 21 of each 28-day cycle and Dexamethasone 40 mg (weekly) and may be reduced to 20 mg (weekly after cycle 6 at the investigator's discretion). Each treatment cycle consists of 28 days.
- Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone: Participants administered with daratumumab 16 mg/kg on Day 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Days 1 and 15 (Cycles 3 to 6), Day 1 (Cycle 7+) along with Lenalidomide 25 mg on Day 1 to 21 of each 28-day cycle and Dexamethasone 40 mg (weekly) and may be reduced to 20 mg (weekly after cycle 6 at the investigator's discretion). Each treatment cycle consists of 28 days.
Period: Overall Study
Arm/Group | Phase 1: 2 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 4 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 8mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone
Started | 3 | 3 | 4 | 3 | 32
Completed | 1 | 2 | 0 | 2 | 16
Not Completed | 2 | 1 | 4 | 1 | 16
Not completed — Adverse Event | 1 | 0 | 3 | 0 | 4
Not completed — Progressive disease | 1 | 1 | 1 | 1 | 10
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: 2 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 4 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 8mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 32 | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.7 (12.74) | 62.7 (2.08) | 57.5 (9.68) | 67.3 (10.26) | 59.7 (8.38) | 60.4 (8.57)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 3 | 2 | 4 | 1 | 22 | 32
  Female | 0 | 1 | 0 | 2 | 10 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  Denmark | 2 | 2 | 1 | 1 | 5 | 11
  France | 0 | 0 | 0 | 1 | 6 | 7
  Italy | 0 | 0 | 0 | 0 | 8 | 8
  Netherlands | 0 | 0 | 3 | 0 | 6 | 9
  United Kingdom | 1 | 1 | 0 | 1 | 4 | 7
  United States | 0 | 0 | 0 | 0 | 3 | 3
Stage of Disease [International Staging System (ISS) [Count of Participants; unit: Participants] — The International Staging System (ISS) system consists of stage I: beta2 microglobulin less than (<)3.5 milligram per liter (mg/L) and albumin greater than or equal to (>=) 3.5 gram/ deciliter (dL) or (35 gram/L); stage II: neither stage I nor stage III and stage III: beta2 microglobulin >= 5.5 mg/L.
  Participants
    Stage I | 0 | 1 | 4 | 1 | 15 | 21
    Stage II | 2 | 1 | 0 | 1 | 14 | 18
    Stage III | 1 | 1 | 0 | 1 | 3 | 6
Number of Prior Lines of Therapy [Count of Participants; unit: Participants]
  1 Line | 0 | 0 | 0 | 0 | 15 | 15
  2-3 Lines | 2 | 3 | 3 | 2 | 17 | 27
  >3 Lines | 1 | 0 | 1 | 1 | 0 | 3
Refractory to Proteasome Inhibitor (PI)/ Immunomodulatory drug (IMiD) [Count of Participants; unit: Participants]
  Both a PI and IMiD | 0 | 0 | 3 | 1 | 0 | 4
  PI only | 0 | 2 | 0 | 0 | 5 | 7
  IMiD only | 0 | 1 | 0 | 1 | 1 | 3
  None | 3 | 0 | 1 | 1 | 26 | 31

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Percentage of Participants With Overall Response Rate (ORR)
Description: ORR is defined as percentage of participants who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR). International Myeloma Working Group (IMWG) criteria (2011)- CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and less than (<) 5 percentage (%) plasma cells in bone marrow; sCR: CR+Normal free light chain ratio and absence of clonal cells in bone marrow by immunohistochemistry or immuno fluorescence; PR: greater than equal to (>=) 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >= 90 percentage (%) or to <200 mg/24 hours; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hour.
Time Frame: Up to 3 years
Population: All treated analysis set included all enrolled participants who received at least one non-zero dose of any study drug during Phase 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase 1: 2 mg/kg Daratumumab + Lenalidomide and Dexamethasone: Participants administered with daratumumab 2 mg/kg on Day 0 (pre dose infusion), 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Days 1 and 15 (Cycles 3 to 6), Day 1 (Cycle 7+) along with Lenalidomide 25 mg on Day 1 to 21 of each 28-day cycle and Dexamethasone 40 mg (weekly) and may be reduced to 20 mg (weekly after cycle 6 at the investigator's discretion). Each treatment cycle consists of 28 days.
- Phase 1: 8 mg/kg Daratumumab + Lenalidomide and Dexamethasone: Participants administered with daratumumab 8 mg/kg on Day 0 (pre dose infusion), 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Days 1 and 15 (Cycles 3 to 6), Day 1 (Cycle 7+) along with Lenalidomide 25 mg on day 1 to 21 of each 28-day cycle and Dexamethasone 40 mg (weekly) and may be reduced to 20 mg (weekly after cycle 6 at the investigator's discretion). Each treatment cycle consists of 28 days.
- Phase 1: Daratumumab (2-16 mg/kg) + Lenalidomide and Dexamethasone: Participants were administered Daratumumab at escalating doses of 2 mg/kg, 4 mg/kg, 8 mg/kg, or 16 mg/kg on Day 0 (pre dose infusion), 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Day 1 of Cycles 3 to 6, and Day 1 of Cycles 7 and beyond. Each cycle consisted of 28 days. Lenalidomide (25 mg was administered orally once daily on Days 1 to 21 of each 28-day cycle) and Dexamethasone (40 mg weekly) were administered concurrently. Dexamethasone dosage could be reduced to 20 mg weekly after Cycle 6 or at the investigator's discretion. Each treatment cycle consisted of 28 days.
Arm/Group | Phase 1: 2 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 4 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 8 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: Daratumumab (2-16 mg/kg) + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 13
Percentage of participants | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 75.0 [19.4 to 99.4] | 66.7 [9.4 to 99.2] | 85.4 [64.8 to 98.1]

2. Primary Outcome: Phase 2: Percentage of Participants With Overall Response Rate (ORR)
Description: ORR is defined as percentage of participants who achieved stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR). IMWG criteria (2011)- CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and less than (<) 5 percentage (%) plasma cells in bone marrow; sCR: CR+Normal free light chain ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; PR: greater than eqaul to (>=) 50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >= 90 percentage (%) or to <200 mg/24 hours; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-protein plus urine M-protein level <100 mg per 24 hour.
Time Frame: Up to 3 years
Population: Intent-to-Treat (ITT) population analysis set included all enrolled participants who signed the informed consent during Phase 2.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone: Participants administered with daratumumab 16 mg/kg on Day 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Days 1 and 15 (Cycles 3 to 6), Day 1 (Cycle 7+) along with Lenalidomide 25 milligram (mg) on Day 1 to 21 of each 28-day cycle and Dexamethasone 40 mg (weekly) and may be reduced to 20 mg (weekly after cycle 6 at the investigator's discretion). Each treatment cycle consists of 28 days.
Arm/Group | Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 32
Percentage of participants | 81.3 [63.6 to 92.8]

3. Secondary Outcome: Phase 2: Duration of Response
Description: Duration of response was calculated from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria (2011).
Time Frame: Up to 5 years
Population: Responders in Intent-to-Treat (ITT) population analysis set included. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 26
Months | NA [26.5 to NA] — Median and the upper bound of the 95% confidence interval (CI) were not estimable due to insufficient number of participants and/or events.

4. Secondary Outcome: Phase 1: Time to Response
Description: Time to first response was defined as the time from the date of first dose of daratumumab to the date of initial documentation of a response (PR or better). Time to best response was defined as the time between the date of first dose of daratumumab and the date of the initial evaluation of the best response (PR or better) to treatment.
Time Frame: Up to 5 years
Population: Responders in all treated population analysis set included. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 1: 2 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 4 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 8 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 3 | 3 | 3 | 2
Months
  Time to first response | 0.99 [0.5 to 1.0] | 1.02 [0.5 to 1.9] | 1.02 [1.0 to 1.8] | 2.25 [1.9 to 2.6]
  Time to best response | 1.9 [1.0 to 6.5] | 13.17 [3.7 to 20.7] | 8.41 [1.0 to 19.9] | 16.72 [6.5 to 26.9]

5. Secondary Outcome: Phase 2: Time to Response
Description: as for outcome 4
Time Frame: Up to 5 years
Population: ITT population analysis set included all enrolled participants who signed the informed consent during Phase 2. Here, 'N' (overall number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 26
Months
  Time to first response | 0.99 [0.5 to 5.6]
  Time to best response | 6.95 [0.5 to 26.8]

6. Secondary Outcome: Phase 2: Time to Progression (TTP)
Description: TTP was defined as the number of days from the date of first infusion (Day 1) to the date of first record of disease progression. Disease progression (IMWG criteria 2011): increase of >=25 percent (%) from lowest response level in Serum M-component and/or (the absolute increase must be >=0.5 g/dL) Urine M-component and/or (the absolute increase must be >=200 mg/24 hour; only in participants without measurable serum and urine M-protein levels: the difference between involved and uninvolved free light chain levels. The absolute increase must be >10 mg/dL; Bone marrow plasma cell percentage: the absolute % must be >=10 %; Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia (corrected serum calcium >11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder. Median TTP was estimated by using the Kaplan-Meier method.
Time Frame: Up to 5 years
Population: ITT population analysis set included all enrolled participants who signed the informed consent during Phase 2.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 32
Months | NA [27.0 to NA] — Median and the upper bound of the 95% CI were not estimable due to insufficient number of participants and/or events.

7. Secondary Outcome: Phase 2: Progression-Free Survival (PFS)
Description: Progression free survival (PFS) was defined as the time between the date of first dose of daratumumab and either disease progression or death, whichever occurs first.
Time Frame: Up to 5 years
Population: ITT population analysis set included all enrolled participants who signed the informed consent during Phase 2.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 32
Months | NA [16.62 to NA] — Median and the upper bound of the 95% CI were not estimable due to insufficient number of participants and/or events.

8. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the number of days from administration of the first infusion (Day 1) to date of death. Median Overall Survival was estimated by using the Kaplan Meier method.
Time Frame: Up to 5 years
Population: ITT population analysis set included all enrolled participants who signed the informed consent during Phase 2.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone
Number analyzed (Participants) | 32
Months | NA [32.23 to NA] — Median and the upper bound of the 95% CI were not estimable due to insufficient number of participants and/or events.

ADVERSE EVENTS:
Time Frame: Deaths: From screening (Day -21) up to 5 years; Serious and Other AEs: From Day 1 up to 50.4 months
Description: All treated analysis set included all enrolled participants who received at least one non-zero dose of any study drug during Phase 1. The safety analysis set included all enrolled participants who received at least one non-zero dose of any study drug during Phase 2.
Groups:
- Phase 1: 2 mg/kg Daratumumab + Lenalidomide and Dexamethasone: Participants received daratumumab 2 mg/kg on Day 0 (pre dose infusion), 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Days 1 and 15 (cycles 3 to 6), Day 1 (cycle 7+) along with lenalidomide 25 milligram (mg) on Day 1 to 21 of each 28-day cycle and dexamethasone 40 mg (weekly) and may be reduced to 20 mg (weekly after cycle 6 at the investigator's discretion). Each treatment cycle consists of 28 days.
- Phase 1: 8mg/kg Daratumumab + Lenalidomide and Dexamethasone: Participants received with daratumumab 8 mg/kg on Day 0 (pre dose infusion), 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Days 1 and 15 (cycles 3 to 6), Day 1 (cycle 7+) along with lenalidomide 25 mg on Day 1 to 21 of each 28-day cycle and dexamethasone 40 mg (weekly) and may be reduced to 20 mg (weekly after cycle 6 at the investigator's discretion). Each treatment cycle consists of 28 days.
- Phase 1: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone: Participants administered with daratumumab 16 mg/kg on Day 0 (pre dose infusion), 1, 8, 15, 22 (cycle 1), Days 1, 8, 15, and 22 (cycle 2), Days 1 and 15 (Cycles 3 to 6), Day 1 (Cycle 7+) along with Lenalidomide 25 milligram (mg) on Day 1 to 21 of each 28-day cycle and Dexamethasone 40 mg (weekly) and may be reduced to 20 mg (weekly after cycle 6 at the investigator's discretion). Each treatment cycle consists of 28 days.
Arm/Group | Phase 1: 2 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 4 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 8mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 1: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone | Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 1/4 | 0/3 | 1/32
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 3/4 | 2/3 | 22/32
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3 | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 2 mg/kg Daratumumab + Lenalidomide and Dexamethasone (N=3) | Phase 1: 4 mg/kg Daratumumab + Lenalidomide and Dexamethasone (N=3) | Phase 1: 8mg/kg Daratumumab + Lenalidomide and Dexamethasone (N=4) | Phase 1: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone (N=3) | Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone (N=32)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 3
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Steroid Withdrawal Syndrome (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Retinal Artery Thrombosis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 2
Sudden Death (General disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 3
Pneumonia Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Influenza A Virus Test Positive (Investigations) | 0 | 0 | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Epstein-Barr Virus Associated Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 3
Cerebral Infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Laryngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 2 mg/kg Daratumumab + Lenalidomide and Dexamethasone (N=3) | Phase 1: 4 mg/kg Daratumumab + Lenalidomide and Dexamethasone (N=3) | Phase 1: 8mg/kg Daratumumab + Lenalidomide and Dexamethasone (N=4) | Phase 1: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone (N=3) | Phase 2: 16 mg/kg Daratumumab + Lenalidomide and Dexamethasone (N=32)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 1 | 8
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 8
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 5
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 4 | 2 | 29
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 0 | 11
Atrial Fibrillation (Cardiac disorders) | 2 | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Hearing Impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Pituitary-Dependent Cushing's Syndrome (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Steroid Withdrawal Syndrome (Endocrine disorders) | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 3 | 1 | 0 | 3
Glaucoma (Eye disorders) | 0 | 1 | 0 | 0 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 0 | 0 | 2
Retinal Artery Thrombosis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 1 | 0 | 0 | 2
Visual Impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vitreous Detachment (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4
Constipation (Gastrointestinal disorders) | 3 | 3 | 1 | 1 | 7
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 3 | 2 | 18
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Faeces Discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 11
Tongue Blistering (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 5
Application Site Erythema (General disorders) | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 4
Chest Pain (General disorders) | 0 | 1 | 0 | 1 | 0
Facial Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 3 | 1 | 4 | 1 | 13
Inflammation (General disorders) | 0 | 0 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 1 | 0 | 4
Oedema (General disorders) | 1 | 1 | 1 | 1 | 3
Oedema Peripheral (General disorders) | 2 | 0 | 1 | 3 | 8
Pain (General disorders) | 0 | 1 | 0 | 0 | 1
Peripheral Swelling (General disorders) | 0 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 1 | 0 | 9
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 1 | 0 | 0 | 0 | 1
Immune System Disorder (Immune system disorders) | 1 | 1 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 9
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 2 | 0 | 1 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Diarrhoea Infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 4
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Herpes Zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 3
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 1 | 1 | 0 | 0 | 3
Kidney Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Lower Respiratory Tract Infection Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 2 | 3 | 2 | 10
Oral Candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Oral Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 4
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 8
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Tooth Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2 | 2 | 0 | 8
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Viral Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 2 | 0 | 0 | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 2 | 0 | 0 | 3
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood Iron Decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 0 | 0 | 0 | 1
Blood Phosphorus Decreased (Investigations) | 1 | 1 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 0 | 2
C-Reactive Protein Increased (Investigations) | 1 | 1 | 0 | 0 | 1
Creatinine Renal Clearance Decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Electrocardiogram QT Prolonged (Investigations) | 1 | 0 | 1 | 1 | 1
Weight Decreased (Investigations) | 0 | 1 | 0 | 0 | 3
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 8
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 6
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Joint Contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 3 | 15
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 3
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Osteonecrosis of Jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 4
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 2
Dizziness Postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 2
Embolic Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 6
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 1 | 3 | 1 | 7
Post Herpetic Neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Visual Field Defect (Nervous system disorders) | 1 | 1 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1
Depressed Mood (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Disinhibition (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 3 | 0 | 8
Mood Altered (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Allergic Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 16
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 3
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 3
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 4
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 3
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin Fragility (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 10
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-09-29): https://cdn.clinicaltrials.gov/large-docs/29/NCT01615029/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT01615029/SAP_001.pdf